CLINICAL TRIAL: NCT01919502
Title: Feasibility and Acceptability of Using a Semi-quantitative Pregnancy Test to Monitor hCG Levels After Assisted Fertility Treatment
Brief Title: Semi-quantitative Pregnancy Test to Monitor hCG Levels After Assisted Fertility Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 6004
Record Dates: First submitted 2013-08-05; First posted 2013-08-09 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Embryo Transfer; Intrauterine Insemination (IUI)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Semi-quantitative urine pregnancy test (Other): Semi-quantitative urine pregnancy test (Quanti5 Multilevel hCG Pregnancy Test)
  Interventions: Device: Semi-quantitative urine pregnancy test

INTERVENTIONS:
Device: Semi-quantitative urine pregnancy test
  Other Names: Quanti5 Multilevel hCG Pregnancy Test

SUMMARY:
Given the potential of semi-quantitative pregnancy tests as part of assisted fertility care, the investigators would like to document the feasibility and acceptability of a semi-quantitative pregnancy test as an adjunct to or replacement of current monitoring protocols to offer women and health care providers a new choice of diagnostic tools to confirm early pregnancy. The pilot will help us to better understand how this tool complements existing monitoring protocols. If a suitable addition or replacement to repeat blood draws for serum hCG assessment, the SQPT could also contribute to efforts to make assisted fertility treatments more patient-friendly. This study seeks to test this innovation by asking women assigned to perform a Quanti5 Multilevel hCG Pregnancy Test (Athenium Pharmaceuticals, LLC, Nashville, TN) at home on a weekly basis for up to 4 weeks after egg retrieval/embryo transfer or intrauterine insemination.

The investigators hypothesize that the test, which can be used at home by women, will provide confirmation of the presence of a pregnancy compared with standard serum hCG testing because 1) it has sensitivity and specificity that correlates well with serum testing, and 2) it can be used at home and thus earlier to determine presence of hCG.

ELIGIBILITY:
Inclusion Criteria:

* Planning embryo transfer or intrauterine insemination (IUI)
* Agrees to return for a series of follow-up visits
* Willing to follow provider instructions regarding use of at-home pregnancy test
* Has not already participated in this study (each woman can only participate once)
* Able to read and write in English
* Willing to provide an address and/or telephone number to be contacted for purposes of follow-up
* Willing and able to consent to study participation

Exclusion Criteria:

* Does not agree to return for a series of follow-up visits
* Not willing to follow provider instructions regarding use of at-home pregnancy test
* Has already participated in this study (each woman can only participate once)
* Not able to read and write in English
* Not willing to provide an address and/or telephone number to be contacted for purposes of follow-up
* Not willing and able to consent to study participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Proportion of SQPT results that accurately monitor pregnancy | 6 weeks
  Participants will have follow-up visits that include serum hCG testing and ultrasounds to confirm pregnancy. Will be able to compare these results to the results of the at-home pregnancy test.

SECONDARY OUTCOMES:
Feasibility of women using this test at home | 6 weeks
  Feasibility of women using this test at home on their own as a potential future substitute or complement to standard sequential clinic-based visits to monitor pregnancy after embryo transfer or IUI. Forms given to document their results at home will include questions on feasibility. Exit interview will also include questions regarding feasibility.
Acceptability of semi-quantitative pregnancy test | 6 weeks
  Acceptability of using semi-quantitative pregnancy at home instead of tests standard clinic-based monitoring after embryo transfer or IUI. Forms given to document their results at home will include questions on acceptability. Exit interview will also include questions regarding acceptability.
Effectiveness of written instructions and provider's counseling | 6 weeks
  Assess if written instructions and provider's counseling enable women using the semi-quantitative pregnancy test at home to understand how it should be used and to correctly interpret the test result. Forms given to document their results at home will include questions on whether the oral and written instructions helped interpret the results. Exit interview will be conducted to determine how the additional information made the participant feel about conducting the test (i.e. more relaxed, less relaxed, or no difference).

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Westphal, MD, Principal Investigator — Division of Reproductive Endocrinology and Infertility Stanford University School of Medicine; Paul Blumenthal, MD, MPH, Principal Investigator — Dept of Obstetrics and Gynecology, Stanford University, Stanford University School of Medicine; Wendy Sheldon, MPH, MSW, PhD, Principal Investigator — Gynuity Health Projects; Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects
Locations (1):
- Stanford University Medical Center, Palo Alto, California, United States

REFERENCES:
- [Derived] Shochet T, Comstock IA, Ngoc NTN, Westphal LM, Sheldon WR, Loc LT, Blum J, Winikoff B, Blumenthal PD. Results of a pilot study in the U.S. and Vietnam to assess the utility and acceptability of a multi-level pregnancy test (MLPT) for home monitoring of hCG trends after assisted reproduction. BMC Womens Health. 2017 Aug 22;17(1):67. doi: 10.1186/s12905-017-0422-y. PMID 28830483